CLINICAL TRIAL: NCT05313308
Title: BUCCOLAM OROMUCOSAL SOLUTION - Special Drug Use Surveillance
Brief Title: A Survey of Midazolam in People With Status Epilepticus
Status: Recruiting | Type: Observational
Sponsor: Clinigen K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: BUCCOLAM PMS; jRCT2031210712 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Midazolam: Participants will receive a single age-specific dose midazolam oromucosal solution through buccal mucosa upon onset of seizures. Dose will be dependent by age of participants as follows: >= 52 weeks and < 1 year; 2.5 mg/dose of midazolam, for >= 1 year and < 5 years; 5 mg/dose of midazolam, for >= 5 years and < 10 years; 7.5 mg/dose of midazolam, for >= 10 years and < 18 years; 10 mg/dose of midazolam. Participants received interventions as part of routine medical care.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Midazolam oromucosal solution
  Other Names: BUCCOLAM oromucosal solution

SUMMARY:
This study is a survey in Japan of midazolam oromucosal solution used to treat people with status epilepticus. The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related from midazolam oromucosal solution and to check if midazolam oromucosal solution improves symptoms of status epilepticus. During the study, participants with status epilepticus will take midazolam oromucosal solution according to their clinic's standard practice. The study doctors will check for side effects from midazolam for 6 months.

ELIGIBILITY:
Inclusion Criteria

* Participants with non-convulsive status epilepticus
* Participants treated with study drug outside the medical institution
* Participants receiving an additional dose of study drug

Exclusion Criteria Participants have any contraindication to midazolam.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with status epilepticus who received midazolam oromucosal solution
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced At Least One Treatment-Emergent Adverse Event (TEAE) | Up to 24 hours after drug administration
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product. It does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a pharmaceutical product (including an investigational product for a new indication in Japan), whether or not related to the pharmaceutical product.
Number of Participants With Serious Adverse Events | Up to 24 hours after drug administration
  A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Number of Participants With Therapeutic Success | Up to 30 minutes after drug administration
  Therapeutic success is defined as cessation of seizure activity within 10 minutes and sustained absence of seizure activity for 30 minutes following the first dose of midazolam oromucosal solution. Number of participants with therapeutic success will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Clinigen K.K.
Locations (1):
- Clinigen selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://jrct.mhlw.go.jp/latest-detail/jRCT2031210712